CLINICAL TRIAL: NCT03697421
Title: Montefiore Medical Center Healthy Marriage and Relationship Education Program
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other); Metis Associates (Unknown)
Responsible Party: Principal Investigator, Traci Maynigo, Program Director, Montefiore Medical Center
Other Study IDs: 2015-5900
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Parenting; Family Relationships
Keywords: parenting; relationships; relationship education; couples; marriage
MeSH Terms: interventions — Occupational Health Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Local Evaluation: The SHR program intends to serves couples who are over 18 years of age, are in a romantic relationship, and have at least one child (biological or adopted) under the age of 18 residing in the home or are expecting.
  Interventions: Other: Relationship Education; Other: Employment Services

INTERVENTIONS:
Other: Relationship Education — We will provide the following 4 activities: 1) marriage and relationship education [using a modified version of the empirically supported Loving Couples, Loving Children (LCLC); 2) pre-marital education and marriage skills; 3) marriage enhancement and marriage skills for married couples; and 4) divorce reduction and relationship skills.
  All couples will be expected to participate in 24 hours of core relationship education workshops (including parenting education). Since parental financial support represents a core element of family stability, relationship education workshops will address motivation for providing financial support through employment for all couples (employed and unemployed) as well as how to manage conflicts over money. All couples will be invited to supplemental workshops (with couples from other cohorts) on topics of specialized interest, including employment services and financial literacy (i.e. budgeting, debt, etc.).
Other: Employment Services — For couples in need of job search, job retention, and career advancement services, we will provide employment services.

SUMMARY:
The proposed program will flexibly provide an array of relationship promotion activities incorporating case management and job placement/career advancement activities: marriage and relationship education; pre-marital education and marriage skills; marriage enhancement and marriage skills for married couples; and divorce reduction and relationship skills. In addition, our proposed local evaluation will examine factors that might account for the observed impacts of attending relationship education programs (i.e., higher levels of relationship satisfaction), including dosage of workshops, relationship commitment and longevity, and skill learning.

DETAILED DESCRIPTION:
The objective of the proposed evaluation is to delineate those factors and sub-groups that account for the observed impact of HMRE services on the quality of relationships. Specifically, we are interested in investigating the following factors:

1. Commitment: Are couples that are more committed to each other (measured in terms of marital status, duration of relationship, or relationship commitment scale scores) more motivated to attend a greater number of HMRE workshops? Do they actually learn more relationship skills, and report improvements in their relationship quality?
2. Hopefulness: How does hopefulness about the relationship impact outcomes?
3. Dosage: Is attendance at a greater number of workshops related to improvements in relationship satisfaction and relationship quality?
4. Couple characteristics: How are various demographic factors related to observed outcomes?
5. Skill acquisition: How much did couples actually learn during the course of the relationship workshop?

In order to explore these research questions, we will be conducting an evaluation that utilizes pre-and post-survey data and qualitative interview information from participants. This will be a descriptive study and not a random assignment design. Data collection will begin when couples who expressed interest in the program attend a preliminary interview with one of Montefiore's clinical staff on site. The program and study will be explained to the couple and they will be asked to consent to participate. Once consent is gathered, on-site staff will administer measures required by our funders through an online system called nForm, or Information, Family Outcomes, Reporting, and Management. This online system was developed by Mathematica Policy Research, an agency contracted by the Department of Health and Human Services to conduct a Cross-Site evaluation of all grantees who received funding to provide relationship education services. Preliminary demographic information will be collected through surveys completed by participants online through secure web browsing at a Montefiore facility.

ELIGIBILITY:
Inclusion Criteria:

* In a committed relationship
* 18 years or older
* expecting a child or are caring for a child in the home at least 50% of the time (biological, foster, adopted, kinship care, etc.)

Exclusion Criteria:

* Active intimate partner violence and increased risk of intimate partner violence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population is 47% Hispanic and 44% African-American. The income level of the majority of the couples enrolled was at or below 200% of poverty level, and 36% received income from public assistance. The majority of couples we served (72%) had a high school degree or less, and nearly half (49%) of participants were unemployed at program enrollment with many more under-employed. Their average age was 36 years old, including 10% between the ages of 17 and 24. The average duration of marriage for couples in our program was 7 years; however, the range of relationship longevity was quite wide, spanning from newlywed couples married for a few months to couples married for over 30 years. All couples had at least one child under 18 years old living in the home (or were expecting a child), and we estimate that approximately two thirds of families in our program were comprised of at least one partner with a child from a previous relationship.
Sampling Method: Non-Probability Sample
Enrollment: 1029 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Couples Satisfaction Index (CSI-32) | Change from Baseline CSI at 6 months
  Considered the gold standard, this measure detects differences in relationship satisfaction with great precision. It is a 32-item scale, total score range from 0 to 161. Higher scores indicate higher levels of relationship satisfaction. CSI-32 scores falling below 104.5 suggest notable relationship dissatisfaction.
Change in Relationship Hope Scale | Change from Baseline Relationship Hope at 6 months
  This is a newly developed 5-item scale by a major relationship researcher (Alan Hawkins), which has reportedly good psychometric properties. It will allow us to hone in on the level of hopefulness and cynicism among our couples. This is a 5-item scale, scores determined by mean, ranging 1-7. Mean scores less than or equal to 5 suggest low hope.
Change in Maybe I Do? Scale (Commitment) | Change from Baseline Commitment at 6 months
  A 4-item measure of commitment developed by another major relationship research group (Scott Stanley and Howard Markman). This is a 4-item scale, with a total score range 1-20. Low commitment is indicated at a total score of 12 or below.
Change in Assessing Emotions Scale (Emotional Intelligence) | Change from Baseline Emotional Intelligence at 6 months
  Assesses the extent individuals perceive, understand, regulate, and harness emotions adaptively. This is a 33-item self-report inventory focusing on typical emotional intelligence. Scores can range from 33 to 165. Low EI is less than or equal to 115 for females and 108 for males; average EI is 116-145 for females and 109-131 for males; high EI is greater than or equal to 146 for females and 132 for male.
Change Skills Assessment Measure (Skill Acquisition) | Change from Baseline Skills at immediately post intervention and at 6 months
  Assesses whether the individual has/has learned the skills and knowledge taught through the program curriculum. There are two forms of this measure, A and B, each 14 items. Scores are percentages ranging from 0-100%. Higher scores represent a higher outcome.
Adverse Childhood Experiences (ACE) Survey | Halfway through intervention (Week 6 of 12 weeks, or Week 5 of 9 weeks)
  The Adverse Childhood Experience (ACE) Questionnaire is a 10-item self-report measure developed for the ACE study to identify childhood experiences of abuse and neglect. Scores range 0-10. Higher scores suggest worse outcomes.

SECONDARY OUTCOMES:
Information, Family Outcomes, Reporting, and Management (nFORM) Applicant Characteristics | Baseline
  This is a survey developed by the Office of Family Assistance utilized by all grantees participating in the national study, that gathers demographic information regarding participants.
Information, Family Outcomes, Reporting, and Management (nFORM) Pre-Program Survey | At start of intervention (Week 1 of 12 or 9 weeks)
  This is a survey developed by the Office of Family Assistance utilized by all grantees participating in the national study that includes questions regarding relationship satisfaction, financial stability, and parenting.
nformation, Family Outcomes, Reporting, and Management (nFORM) Post-Program Survey | Immediately post intervention (Week 12 of 12 weeks or Week 9 of 9 weeks)
  This is a survey developed by the Office of Family Assistance utilized by all grantees participating in the national study that includes questions regarding relationship satisfaction, financial stability, and parenting.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wetzler, PhD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No